CLINICAL TRIAL: NCT01279837
Title: Muscle Preservation and Swallow Function Following Radiotherapy: A Dose Response Study
Brief Title: Pharyngocise Dose Response Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: RSG-06-103-01(CCE)
Record Dates: First submitted 2011-01-07; First posted 2011-01-19 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2011-01

CONDITIONS: Dysphagia
Keywords: swallowing disorders; swallowing therapy; head neck cancer; oropharyngeal dysphagia
MeSH Terms: conditions — Deglutition Disorders; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual care (No Intervention): Control (Usual care) group in which patients will receive swallowing and prescribed dietary intervention during the radiotherapy period prescribed by the attending physician.
- High Intensity Pharyngocise (Experimental): Patients receive twice daily swallowing intervention by a speech language pathologist, consisting of the battery of isometric / isotonic exercises.
  Interventions: Behavioral: Pharyngocise
- Low Intensity Pharyngocise (Active Comparator): Patients will receive a one time only swallowing intervention session by a speech language pathologist, instructing them in the battery of isometric / isotonic exercises plus a home practice instruction digital video tape to support self directed practice of this program at home.
  Interventions: Behavioral: Pharyngocise

INTERVENTIONS:
Behavioral: Pharyngocise — swallowing intervention by a speech language pathologist, consisting of the battery of isometric / isotonic exercises
  Arms: High Intensity Pharyngocise; Low Intensity Pharyngocise

SUMMARY:
In this study supported by an American Cancer Society grant, the investigators are evaluating two levels of swallowing exercise intensity on the maintenance of swallowing muscles and their function in Head/Neck cancer patients undergoing radiotherapy. Patients in this study are randomly placed into different exercise groups and provided with exercises to perform daily during their radiation treatment. Their progress, diet management and swallowing ability are monitored throughout the treatment period and followed up until 3 months after radiation treatment. In addition to the daily treatment details, the patients perception of their swallowing ability and concerns about their health and treatment are also measured. This clinical trial will help to refine a previously investigated simple exercise package and provide a program of intervention that can help prevent medically related complications of swallowing difficulty (e.g. pneumonia, dehydration, prolonged tube feeding), and improve the ability to eat for patients with head / neck cancer. Ultimately it is hoped that this form of exercise therapy will help reduce the costs (personal and financial) to the patient, caregivers and community.

DETAILED DESCRIPTION:
In an earlier pilot study, a regime of simple swallowing exercises was identified as useful in maintaining oropharyngeal muscle characteristics as measured by T2 weighted Magnetic Resonance Imaging (MRI) and produced a trend toward improved function for swallowing in patients undergoing radiotherapy for head and neck cancer. The purpose of this current study is to evaluate the dose response of two levels of swallowing exercise intensity on the maintenance of muscle composition and function for swallowing in Head/Neck cancer patients undergoing radiotherapy.

HYPOTHESIS: A program of intensive swallowing exercise (Pharyngocise) will maintain muscle function in the oral cavity and pharynx during radiotherapy, preserving or supporting swallowing function in Head/Neck cancer patients.

STUDY DESIGN: 130 patients with Head/Neck cancer, confirmed by clinical history and exam, will be recruited over a 4 year period. All subjects will undergo an initial baseline work up, including a standardized clinical and instrumental swallowing evaluation, psychosocial scales, nutritional exam, and T2 weighted MRI prior to the first radiation therapy. Subjects will be randomized into 1 of 3 groups:

Group A: Usual care (control) group - patients will receive swallowing and prescribed dietary intervention during the radiotherapy period prescribed by the attending physician.

Group B: High intensity pharyngocise treatment group - patients will receive twice daily swallowing intervention by a speech language pathologist, consisting of the battery of isometric/isotonic exercises.

Group C: Low intensity pharyngocise treatment group - patients will receive a single instructional exercise session on the isometric/isotonic exercises from a Speech Language Pathologist and a practice tape to support home practice of the exercises.

All patients will be treated for approximately 6 weeks and followed for 3 months post treatment. Baseline assessments will be repeated. In addition, daily treatment details, patients perception of current swallowing ability and progress in therapy will be recorded by the Speech Pathologist. Participants will be independently monitored throughout the treatment period by researcher blind to the treatment group assigned, via weekly phone interview sessions. Compliance with the treatment techniques, and the occurrence of any negative endpoints such as occurrence of aspiration pneumonia will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Head/Neck cancer of the oropharyngeal or adjacent regions, confirmed by clinical history and exam, with positive cross sectional imaging studies and histopathological biopsy excluding other pathology.
2. Planned external beam radiation therapy
3. No previous history of non-oral feeding for cancer related illness
4. Able to undergo MRI imaging scan
5. Patient and physician agreement to enter the study

Exclusion Criteria:

1. Planned extensive surgical intervention
2. Existence of a co-existing neurological or medical disorder known to cause dysphagia
3. Prior radiotherapy or surgery to the head / neck region that could contribute to dysphagia.
4. Previous swallowing therapy within four weeks of randomization
5. Gross tumor involvement of the oral and pharyngeal muscles obviating adequate MRI measurements of the majority of muscles of interest.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-06; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Change in T2 Weighted Magnetic Resonance Imaging | at 3 months after treatment
  T2 Weighted Magnetic Resonance Imaging (MRI) to quantify baseline muscle parameters in the oral cavity and pharynx. The regions of interest will be identified on images using axial and coronal planes. Information regarding the muscle volume, composition (fat Vs muscle Vs edema) as reflected by the signal intensity.
Clinical swallowing Ability | baseline, 3 weeks, 6 weeks and 3 months post treatment
  Swallowing ability and method/ type of dietary intake, e.g. Functional Oral Intake Scale score [F.O.I.S] over the study period

SECONDARY OUTCOMES:
Weight | baseline, 3 weeks, 6 weeks and 3 months post treatment
  Weight and Body Mass Index will be calculated.
Psychosocial functioning | baseline and 3 months post treatment
  Domain assessments for, quality of life, pain,and fatigue using the Functional Assessment of Cancer Therapy - Head and Neck (FACT-H/N), Pain Disability Index (PDI), Functional Assessment of Cancer Therapy - Anemia (FACT-An) scale, Multidimensional Fatigue Symptom Inventory (MFSI), Profiles of Mood Scale (POMS) and Center for Epidemiologic Studies Depression Scale(CESD).
Instrumental swallowing evaluation | baseline and 3 months post treatment
  Range of swallowing biomechanics measured from endoscopic and fluorographic evaluations.
Swallowing Quality of Life | baseline and 3 months post treatment
  Patient perception of effect of swallowing disability - Swallowing Quality of Life (SWAL QOL) score during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Giselle Carnaby-Mann, PhD, Principal Investigator — University of Florida
Locations (1):
- Shands Cancer Center, University of Florida, Gainesville, Florida, United States